CLINICAL TRIAL: NCT02878668
Title: The Predictor of Infectious Complication After Hepatopancreatobiliary Surgery and Monitoring Indicator of Anti-infectious Therapy
Brief Title: The Value of Infectious Biomarkers for Prediction of Complication After Hepatopancreatobiliary Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Changhai Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); West China Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); First Affiliated Hospital of Harbin Medical University (Other); Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Wenhui Lou, professor, Shanghai Zhongshan Hospital
Other Study IDs: ZS-LWH-2016
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Post-operative Complication
Keywords: procalcitonin; post-operative; complication; CRP

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: hepatopancreatobiliary surgery — hepatopancreatobiliary surgery

SUMMARY:
Post operative complication after hepatopancreatobiliary surgery is high as 30-50%，which is the main reason for patient admitted to ICU. Several biomarkers have been shown to be useful in the early diagnosis of sepsis and systemic bacterial infection. The purpose of this study is to assess the predictive value of biomarkers for early complication after hepatopancreatobiliary surgery and assess the effectiveness of anti-infectious therapy.

DETAILED DESCRIPTION:
Postoperative complication after major abdominal surgery, such as pancreatic surgery and hilar cholangiocarcinoma surgery, is higher, up to 30 to 50%.It is the mainly reason for the patient to admit to ICU. Among this, the most common and difficult to handle complication is mainly anastomotic fistula, abdominal effusion and subsequent secondary infection. Delayed diagnosis can cause systemic inflammatory response syndrome (SIRS), multiple organ failure ( MODS), and even death. From a surgical point of view, it leads to surgical failure and often need the second surgery. However, the diagnosis and treatment of postoperative infection is also facing two problems: it is difficult to confirm the diagnosis and make treatment decision. Hence, there is a strong need of an additional tool to early diagnose post operative complication.

Serum procalcitonin (PCT), is a 116 amino-acids protein produced by C-cells of the thyroid gland. PCT baseline levels are low (<0.05 ng/ml), but increase significantly in patients with severe bacterial infections. Therefore, PCT levels are used to monitor the course and prognosis of systemic bacterial infections and to tailor the therapeutic interventions more efficiently. Furthermore, PCT could serve as an early predictive marker for the clinical course of septic complications after abdominal surgery. The aim of this study is to demonstrate if PCT is a more sensible, specific and reliable biomarker of post operative complication than other biomarkers

The investigators conducted a observational, prospective study. All patients undergoing electively hepatopancreatobiliary surgery in seven centres are recruited. In all cases white blood count (WBC), C-reactive protein (CRP) and PCT levels are measured in 1st, 3rd and 5th postoperative day (POD). Informed consent was obtained in all patients.The study is approved by the hospital's Ethical Committee.

ELIGIBILITY:
Inclusion Criteria:

* age > = 18 years
* Hospitalized patients with elective hepatopancreatobiliary surgery

Exclusion Criteria:

* age <18 years
* emergency operative patients
* Preoperative fever, white blood cell elevation and preoperative infection
* Systemic inflammatory disease
* renal failure
* hematology disease
* preoperative abnormal PCT, IL-6, IL-8, CRP
* Laparoscopic cholecystectomy
* Bile duct infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000 elective hepatopancreatobiliary sugery hospitalized patients will be included
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
post operative complication | within the first 30 days after he operation

SECONDARY OUTCOMES:
sepsis | within the first 30 days after he operation

CONTACTS AND LOCATIONS:
Overall Officials: Wenhui Lou, MD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (7):
- China (7):
  - Beijing Friendship hospital, Capital Medical University, Beijing, Beijing Municipality
  - Sun Yat-Sen Memorial Hospital，Sun Yat-Sen University, Guangzhou, Guangdong
  - The first affiliated hospital of Harbin Medical University, Harbin, Heilongjiang
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Assicot M, Gendrel D, Carsin H, Raymond J, Guilbaud J, Bohuon C. High serum procalcitonin concentrations in patients with sepsis and infection. Lancet. 1993 Feb 27;341(8844):515-8. doi: 10.1016/0140-6736(93)90277-n. PMID 8094770
- [Background] Mofidi R, Suttie SA, Patil PV, Ogston S, Parks RW. The value of procalcitonin at predicting the severity of acute pancreatitis and development of infected pancreatic necrosis: systematic review. Surgery. 2009 Jul;146(1):72-81. doi: 10.1016/j.surg.2009.02.013. Epub 2009 May 8. PMID 19541012
- [Background] Rau BM, Frigerio I, Buchler MW, Wegscheider K, Bassi C, Puolakkainen PA, Beger HG, Schilling MK. Evaluation of procalcitonin for predicting septic multiorgan failure and overall prognosis in secondary peritonitis: a prospective, international multicenter study. Arch Surg. 2007 Feb;142(2):134-42. doi: 10.1001/archsurg.142.2.134. PMID 17309964
- [Background] Novotny AR, Emmanuel K, Hueser N, Knebel C, Kriner M, Ulm K, Bartels H, Siewert JR, Holzmann B. Procalcitonin ratio indicates successful surgical treatment of abdominal sepsis. Surgery. 2009 Jan;145(1):20-6. doi: 10.1016/j.surg.2008.08.009. Epub 2008 Sep 26. PMID 19081471
- [Background] Limper M, de Kruif MD, Duits AJ, Brandjes DP, van Gorp EC. The diagnostic role of procalcitonin and other biomarkers in discriminating infectious from non-infectious fever. J Infect. 2010 Jun;60(6):409-16. doi: 10.1016/j.jinf.2010.03.016. Epub 2010 Mar 27. PMID 20347867
- [Background] Tavares E, Maldonado R, Ojeda ML, Minano FJ. Circulating inflammatory mediators during start of fever in differential diagnosis of gram-negative and gram-positive infections in leukopenic rats. Clin Diagn Lab Immunol. 2005 Sep;12(9):1085-93. doi: 10.1128/CDLI.12.9.1085-1093.2005. PMID 16148175
- [Background] Scapini P, Lapinet-Vera JA, Gasperini S, Calzetti F, Bazzoni F, Cassatella MA. The neutrophil as a cellular source of chemokines. Immunol Rev. 2000 Oct;177:195-203. doi: 10.1034/j.1600-065x.2000.17706.x. PMID 11138776
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] DeOliveira ML, Winter JM, Schafer M, Cunningham SC, Cameron JL, Yeo CJ, Clavien PA. Assessment of complications after pancreatic surgery: A novel grading system applied to 633 patients undergoing pancreaticoduodenectomy. Ann Surg. 2006 Dec;244(6):931-7; discussion 937-9. doi: 10.1097/01.sla.0000246856.03918.9a. PMID 17122618
- [Background] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309